CLINICAL TRIAL: NCT05531903
Title: High-density Activation Mapping of the Slow Pathway During Sinus Rhythm: a New and Simple Method to Guide Catheter Ablation in Patients With Typical Atrioventricular Nodal Reentrant Tachycardia
Brief Title: High-density Activation Mapping of the Slow Pathwayto Guide Catheter Ablation in Patients With Typical Atrioventricular Nodal Reentrant Tachycardia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Jesus Ignacio Jimenez Lopez, Principal investigator, Parc de Salut Mar
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEIm 2022/10521
Record Dates: First submitted 2022-08-28; First posted 2022-09-08 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Supraventricular Tachycardia; Atrioventricular Nodal Re Entrant Tachycardia
MeSH Terms: conditions — Tachycardia, Supraventricular; Tachycardia, Atrioventricular Nodal Reentry

STUDY DESIGN:
Intervention Model Description: Single group of intervention. A control group with absence of dual AVN phisiology to check lack of abnormal fragmented/slow conduction confluent zones.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients with atrioventricular node reentrant tachycardia (Experimental): Patient with documented AVNRT and fragmented/slow conduction zones observed in a 3D high density mapping
  Interventions: Device: Description of Slow pathway signals to facilitate ablation

INTERVENTIONS:
Device: Description of Slow pathway signals to facilitate ablation — 3D endocardial mapping in order to identify slow pathway signals and abolish or modificate them after radiofrequency ablation

SUMMARY:
Atrioventricular nodal reentrant tachycardia (AVNRT) is the most common supraventricular tachycardia inducible during an electrophysiological study. Although ablative therapy proved to be the treatment of choice, little is known about the components of the tachycardia circuit. The aim of this study is to detect the presence and patterns of specific electrograms representing slow pathway (SP) potentials and to explore Koch's triangle pattern activation during sinus rhythm and/or atrial extraestimulus with a high-density mapping catheter in an attempt to clarify a fast and safety catheter ablation strategy. We hypothesized that, in patients with dual atrioventricular nodal physiology, during sinus rhythm (SR), high-density mapping (HDM) catheters could identify the SP signals, making possible to delineate small areas of slow conduction associated to abnormal electrograms on Koch's triangle. On a second step, radiofrequency (RF) applications safety guided by the HDM obtained with this method, should interrupt the circuit far from the His region. Finally, SP signals should disappear after the RF procedure when performing a new 3D HDM. A control group of patients without AVN dual physiology should show absence of fragmented/slow conduction zones.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 yo with AVNRT observed after electrophysiological study

Exclusion Criteria:

* Patients < 18 yo

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Absence of reinduction of AVNRT after abolition of fragmented/slow conduction signals | one day
  Number of patients with absence of fragmented/slow conduction signals observed during sinus rhythm or atrial pacing after radiofrequency application

SECONDARY OUTCOMES:
Absence of AVNRT relapses | one month
  Number of patients with absence of relapses after 1 month of the electrophysiological study
Percentage of patient without AVNRT reinduction after procedure | One day
  Percentage of patients without tachycardia induction after radiofrequency applications protocol

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Ignacio Jimenez López, MD, Principal Investigator — Parc de Salut Mar
Locations (1):
- Jesús Ignacio Jiménez López, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be register with RED CAP